CLINICAL TRIAL: NCT02571465
Title: Assessment of Fluid Responsiveness in Patients After Cardiac Surgery Comparison of Different Functional Hemodynamic Parameters and Tests
Brief Title: Assessment of Fluid Responsiveness in Patients After Cardiac Surgery
Acronym: POP
Status: Completed | Type: Observational
Sponsor: Triemli Hospital (Other)
Responsible Party: Principal Investigator, Christoph K Hofer, MD DEAA, Triemli Hospital
Other Study IDs: IFA10-3
Record Dates: First submitted 2015-10-07; First posted 2015-10-08 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Hemodynamics; Patient Monitoring
Keywords: functional hemodynamic parameter; passive leg raising; stroke volume variation; pulse pressure variation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Passive leg raising test and fluid challenge

SUMMARY:
To overcome the limited accuracy of functional hemodynamic parameters such as stroke volume and pulse pressure variation (SVV and PPV) during spontaneous breathing, a Passive Leg Raising (PLR) manoeuvre has been suggested as a reliable predictor of fluid responsiveness.

Aim of this study was to evaluate fluid responsiveness using SVV, PPV and PLR during the transition from controlled to spontaneous breathing in cardiac surgery patients

DETAILED DESCRIPTION:
In patients after elective off-pump CABG are enrolled hemodynamic measurements are performed in the postoperative period upon arrival in the ICU using a PiCCO2 system (Pulsion Medical Systems, Munich, Germany).

Controlled fluid challenges (500 ml) are done at 3 time-points:

A) during controlled mechanical ventilation B) during pressure support ventilation with spontaneous breathing and C) after extubation.

Stroke volume (SV), SVV and PPV as well as standard hemodynamic parameters (MAP = mean arterial pressure, HR = heart rate) are assessed.

A PLR is performed before fluid administration at all 3 time points. A positive response is defined as an increase in SV>15 %.

Prediction of fluid responsiveness will be tested by AUC (area under the receiver operating characteristic - ROC - curve).

ELIGIBILITY:
Inclusion Criteria:

* preserved left ventricular function
* regular heart rhythm

Exclusion Criteria:

* emergency procedures
* intra- and extra-cardial shunts
* aortic and tricuspid valve insufficiencies
* peripheral arterial occlusive disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective off-pump CABG
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-04; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Stroke volume increase > 15% | 20 min
  Stroke volume increase defines fluid responsiveness

CONTACTS AND LOCATIONS:
Overall Officials: Christoph K Hofer, MD DEAA, Principal Investigator — Triemli City Hospital
Locations (1):
- Triemli City Hospital, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Marik PE, Cavallazzi R, Vasu T, Hirani A. Dynamic changes in arterial waveform derived variables and fluid responsiveness in mechanically ventilated patients: a systematic review of the literature. Crit Care Med. 2009 Sep;37(9):2642-7. doi: 10.1097/CCM.0b013e3181a590da. PMID 19602972
- [Background] Monnet X, Rienzo M, Osman D, Anguel N, Richard C, Pinsky MR, Teboul JL. Passive leg raising predicts fluid responsiveness in the critically ill. Crit Care Med. 2006 May;34(5):1402-7. doi: 10.1097/01.CCM.0000215453.11735.06. PMID 16540963
- [Derived] Ganter MT, Geisen M, Hartnack S, Dzemali O, Hofer CK. Prediction of fluid responsiveness in mechanically ventilated cardiac surgical patients: the performance of seven different functional hemodynamic parameters. BMC Anesthesiol. 2018 May 22;18(1):55. doi: 10.1186/s12871-018-0520-x. PMID 29788919